CLINICAL TRIAL: NCT04040101
Title: Development of a Smartphone-based Balance Assessment System for Subjects With Chronic Stroke
Brief Title: Smartphone-based Balance Assessment System for Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-107-05-048
Record Dates: First submitted 2019-07-14; First posted 2019-07-31 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Adult (No Intervention): balance assessment
- Stroke (No Intervention): balance assessment
- Stroke smartphone training (Experimental): smartphone balance training
  Interventions: Device: smartphone-based balance training system
- Stroke traditional training (Active Comparator): traditional physical therapy training
  Interventions: Device: smartphone-based balance training system

INTERVENTIONS:
Device: smartphone-based balance training system — use smartphone application to training balance
  Other Names: traditional physical therapy
  Arms: Stroke smartphone training; Stroke traditional training

SUMMARY:
Background:

Stroke is the 4th deadly disease in Taiwan, 2016. Long term disabilities, balance impairments and limitations of activities of daily living are common characteristics of stroke. Balance assessment and training play an important role in stroke rehabilitation. However, there are some limitations. Clinical assessments (functional scales) could not avoid some errors caused by subjective observations from different test givers; instrumental assessments (force plates, Biodex system) are complex to approach, not easy to use, and difficult to get. Balance training could not meet the expected effectiveness due to inconvenient transportations, forgotten home programs, and time limitation caused by huge amount of patients with insufficient therapists. Smartphones had been used for health promoting and sport training. The balance training related applications could be found at Google Play store, but clinically proved effective App and stroke-designed App has not yet existed. The balance rehabilitation of stroke sufferers will be benefited if there is an easy-use and effective App that supports balance assessment and personalized training by combining the convenience and powerfulness of smartphones.

Purpose:

The purposes of this study are: Year 1 Develop a smartphone-based application to assess and train static balance for stroke sufferers, and evaluate the feasibility of the application; Year 2 Develop a smartphone-based application to assess and train dynamic balance for stroke sufferers, and evaluate the feasibility of the application; Year 3 Build a static and dynamic balance performance standard by recruiting healthy subjects, then evaluate the training effects of the application on balance performance of stroke sufferers.

Methods:

Android smartphones will be used to analyze the balance performance by collecting acceleration and angular velocity data from the built-in sensors. Static balance assessment and training system will be developed in the first year. The system will assess balance ability by testing the performance under different standing conditions, then provide a training plan according to the assessment result. Dynamic balance assessment and training system will be developed in the second year. The system will execute limits of stability test to assess dynamic balance, then provide a training plan according to the assessment result. Validity and reliability will be tested in the first and second year, by comparing the smartphone assessment result with Berg balance scale, force plate, and Biodex balance system. In the third year, we will recruit healthy subjects to create a balance performance standard, then recruit chronic stroke subjects to evaluate the training effect of the App by comparing with traditional rehabilitation therapy.

Expected Results & Contribution When the study is completed, several valuable contributions will be provided. These include (1) developing a smartphone application which can be used to assess and rehabilitate static and dynamic balance functions on stroke sufferers; (2) evaluating the feasibility and the training effects of the smartphone application, and providing evidence-based results for scientific paper publication; (3) clinically offering an easy-used and effective tool for clinicians and subjects with stroke to evaluate and improve balance performance.

ELIGIBILITY:
Inclusion Criteria:

* stroke
* Brunnstrom stage > 4
* able to walk independently indoors
* able to follow order of the researchers

Exclusion Criteria:

* have any diseases that may affect balance performance except stroke

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Balance performance assessed by smartphone-based balance test | 4 weeks
  The data of smartphone built-in accelerometer and gyroscope will be measured and calculated
Balance performance assessed by force plates | 4 weeks
  The movement of center of pressure (COP) will be measured and calculated
Balance performance assessed by Berg balance scale | 4 weeks
  The score of Berg balance scale will be measured

CONTACTS AND LOCATIONS:
Overall Officials: You-Ruei Hou, Master, Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: No